CLINICAL TRIAL: NCT02297919
Title: Eskisehir Osmangazi University- Scientific Research Projects
Brief Title: Evaluation of the Effectiveness of Internet Based Nutrition and Physical Activity Education Programme in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Fatih Oz, Public Health, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 80558721/244
Record Dates: First submitted 2014-11-06; First posted 2014-11-21 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Obesity
Keywords: Web-based education, Adolescent, Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- web based intervention (Experimental): Web based intervention: Students will have access to the educational content through the learning management system on the web site (genc-e-saglik) created for this project.
  Interventions: Behavioral: Effectiveness of Internet Based Obesity Control Programme
- classic preprepared lesson (Active Comparator): Training at the control group,lectures will be presented on the basis of the classic preprepared lesson by educator and at the end of the training, will be answered student's questions.
  Interventions: Behavioral: Effectiveness of Internet Based Obesity Control Programme

INTERVENTIONS:
Behavioral: Effectiveness of Internet Based Obesity Control Programme

SUMMARY:
The purpose of this study to create an educational portal "Genç (e) sağlık" in an attempt to develop a healthy eating habit, increase physical activity and reduce sedentary behavior in order to prevent to overweight gain which is school-based approach in adolescents and there with also test the level of program information and the behavioral alterations of effectiveness.

DETAILED DESCRIPTION:
This interventional study was planned to be conducted on high school class 1 students from the city center of Eskisehir. With considering a method success of 40%, thenew approach is expected to increase the success rate to 55%. In this study that will be carried out on two sets of methods, the sample size needed is estimated to be 175 individual with 95% confidence and 80% power.

Because of the three-stage nature of the study and characteristics of study population, it was planned to include approximately 250 students in each group with raising the estimated sample size by 50%. There are 3 high schools (Ahmet Kanatli Anatolian High school, Kilicoglu Anatolian High school and Ahmet Yesevi Anatolian High school) with an established internet infrastructure which were included in the Fatih Project implemented by the Ministry of Education and tablet PCs were provided to the students studying these three schools in Eskisehir.

Tablet PCs were only provided to the class 1 students. A total of 550 students getting education and training in these 18 class 1 classrooms in these three school were planned to be included in the study. Of the classrooms, 9 were considered to be randomized as interventional group and other 9 were as control groups.

After obtaining the necessary permissions to perform the study, measured body weights and heights of all students and calculated body mass index and physical activiti evaluated by pedometre. Number of steps will be measured with the pedometer at the beginning and at the end of the week all students. Conduct a questionnaire, which is accepted in the international literature, the School Physical Activity and Nutrition(SPAN) has been modified and validated Turkish version of questionnaire will be applied.

Students will have access to the educational content through the learning management system on the web site (genç-e-saglık) created for this project. The images and links appropriate to the age of the students will be present in the home page. There will be 4 parts consisting of a Myself assessments (to provide individual feedback to the user), a communication channel through which students can ask relevant questions, a media offering the weekly content of the courses, as well as another part including a variety of interactions and fun games. Weekly courses will include a total of 4 lessons, with 2 lessons on nutrition and one each lessons on obesity and physical activity. Each lesson was planned to take approximately 15 minutes. A short assessment form including 5 questions will be included at the end of each course and it will be designed to inform the students how many right answers they gave at the end of the test. The program is scheduled to continue for 4 months. During the each training period, will be send a letter for family and a CD which is recorded the training program. Besides that submit a claim to sign and send back a document that they have committed to participate in the program and time spent towatch CD. Training at the control group,lectures will be presented on the basis of the classic preprepared lesson by educatorand at the end of the training, will be answered student's questions. Before and after the training, will be considered to survey the level of knowledge by questions. After the completion of the four monthly training program, at the sixth month of study, will be evaluated to the height and weight measurement, determination of the number of steps and the latest state of students by SPAN questionnaire physical activiti evaluated by pedometre. At the end of the study, an assembly will be arranged to given gifts to participating schools, students which is participating in all phases of the study and who achieved success evaluation of the level of knowledge more over presented the results of the project.

ELIGIBILITY:
Inclusion Criteria:

* All students who accept to participate in the study

Exclusion Criteria:

* Students who refused to participate in the study

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Eating habit and behaviour will assess. The height and weight of student's will measure. | four months

CONTACTS AND LOCATIONS:
Overall Officials: Selma Metintas, Study Director — Eskisehir Osmangazi University Medicine Faculty Department of Public Health
Locations (1):
- Eskisehir Osmangazi University Medicine Faculty Department of Public Health, Eskişehir, Turkey (Türkiye)